CLINICAL TRIAL: NCT00048763
Title: Safety and Efficacy of Pletal(Cilostazol) for the Treatment of Juvenile Primary and Secondary Raynaud's Phenomenon
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Otsuka America Pharmaceutical (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 21-01-335
Record Dates: First submitted 2002-11-07; First posted 2002-11-11 (Estimated); Last update posted 2005-07-19 (Estimated); Status verified 2005-07

CONDITIONS: Raynaud's Disease
Keywords: circulatory; vascular; idiopathic
MeSH Terms: conditions — Raynaud Disease | interventions — Cilostazol

INTERVENTIONS:
Drug: Pletal

SUMMARY:
Juvenile primary Raynaud's (ray-knows) Phenomenon is a disorder of the blood vessels in the fingers and sometimes can affect the toes, nose, or ears. When children with primary Raynaud's Phenomenon are exposed to chilly or cold conditions from weather, cold temperatures, or even holding cold items from the refrigerator, their fingers may become cold, numb, hurt, and/or turn purple or white. Children with primary Raynaud's Phenomenon have no underlying systemic disease. The cause for their symptoms is unknown. The investigational drug, Pletal(cilostazol), which has been approved for other conditions, inhibits the ability of one type of blood cell, platelets, to form blood clots, and also widens narrowed blood vessels. It has been used in a variety of other conditions in which blood flow is decreased. This study will test the safety and effectiveness Pletal(cilostazol) to lessen the severity of the symptoms and decrease the number of primary Raynaud's episodes in juvenile patients.

ELIGIBILITY:
Inclusion critera:

* 5 to 6 years old
* fulfill diagnostic criteria for primary or secondary Raynaud's

Ages: 5 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 75
Dates: Start 2001-10; Study Completion 2003-06

CONTACTS AND LOCATIONS:
Locations (18):
- United States (18):
  - Advanced Medical Clinical Therapeutics, Anchorage, Alaska
  - Advanced Medical Research Institute, Fresno, California
  - Madera Family Medical Group, Madera, California
  - Connecticut Children's Medical Center, Hartford, Connecticut
  - LaRabida Children's Hospital, Chicago, Illinois
  - Children's Hospital Boston, Boston, Massachusetts
  - St. Louis University Health Sciences Center, St Louis, Missouri
  - Children's Hospital, Omaha, Nebraska
  - Asthma & Allergy Research Center, Newark, New Jersey
  - SUNY Downstate Medical Center, Brooklyn, New York
  - Children's Hospital of Buffalo, Buffalo, New York
  - Schneider Children's Hospital, New Hyde Park, New York
  - New York Medical College, Valhalla, New York
  - Jobst Vascular Center, Toledo, Ohio
  - The Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Monarch Research Associates, Norfolk, Virginia
  - Children's Hospital and Regional Medical Center, Seattle, Washington